CLINICAL TRIAL: NCT03534999
Title: Effect of Transcutaneous Electrical Nerve Stimulation on Pain Intensity of Patients With Hip Arthroplasty: A Randomized Control Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation on Pain Intensity of Patients With Hip Arthroplasty
Acronym: TENSHIParth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obafemi Awolowo University (Other)
Responsible Party: Principal Investigator, Adesola Ojo Ojoawo, Principal Investigator, Obafemi Awolowo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OJO/2018/002
Record Dates: First submitted 2018-04-30; First posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Hip Fractures
Keywords: TENS,; VAS,; Oxford-Hip-score,; Hip-arthroplasthy,; Pain-intensity
MeSH Terms: conditions — Hip Fractures; Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Patients with Hip Arthroplasty, one group was on TENS other group was a control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Experimental): This is intervention Group. Patients in this group received Transcutaneous Electrical Nerve Stimulation (TENS). The VAS and Oxford hip score was administered prior to the treatment to ascertain their pain intensity and hip disability level. The site of intervention (5cm away from incision site) was cleaned properly with cotton wool soaked in methylated spirit in an outward motion. Before the self-adhesive, pre gelled electrodes was placed on the cleansed sites.The TENS unit was switched on and the parameters was adjusted to the required level. For this study, parameters used are: 100µs pulse duration, 100Hz frequency and an intensity comfortable for the patient for a duration of 15 minutes.
  Interventions: Device: Experimental. This was the group that received TENS; Other: No intervention
- Control (No Intervention): This was the group with no intervention. Subjects were on their normal analgesic and antibiotic medication for the period of research. The VAS and Oxford hip score were administered on the first day to ascertain pain intensity and hip disability level. The subject continued on the normal analgesics only till the third day and VAS and Oxford hip score was re-administered to assess any change in the pain intensity and hip disability level.

INTERVENTIONS:
Device: Experimental. This was the group that received TENS — Patients that were on TENS . They were treated twice daily for 5 days. VAS and Hip Score scale were used to assess the pain intensity and disability level
  Other Names: TENS
  Arms: TENS
Other: No intervention — Patients in this group were on their drugs only. There was no physiotherapy intervention for the patient. VAS and Hip Score scale were used to ascertain the pain intensity and hip disability at the before the treatment and after the treatment
  Other Names: Control
  Arms: TENS

SUMMARY:
Fifty patients with hip arthroplasty were purposively recruited for the study. They were allocated into two groups randomly with equal number. One group had TEN, other served as control. Pain intensity was measured every day of the treatment.

DETAILED DESCRIPTION:
Subjects that participated were post-surgical patients with hip arthroplasty receiving treatment at Orthopedic Ward of Obafemi Awolowo University Teaching Hospitals Complex (OAUTHC), Ile-Ife. Excluded from the study were subjects who had surgery but have infected wound, those with deep vein thrombosis, and those with thrombophlebitis post-surgery. The subjects were allocated randomly into 2 groups; one group of 25 patients was on TENS (experimental group) and the other group of 25 patients was on their normal drugs without TENS (control group). Before the start of intervention, the procedure of the intervention and the way the subject would feel during the course of the intervention was explained to the subject and the consent of the patient was obtained. The procedure was as follows:The Visual Analogue Scale and Oxford hip score was administered prior to the treatment to ascertain their pain level and hip disability before the treatment. The site of intervention (5cm away from incision site) was cleaned properly with cotton wool soaked in methylated spirit in an outward motion. Before the self-adhesive, pre gelled electrodes was placed on the cleansed sites. The TENS unit was switched on and the parameters was adjusted to the required. For this study, parameters used are: 100µs pulse duration, 100Hz frequency and an intensity comfortable for the patient for a duration of 15 minutes.

At the expiration of treatment, the electrodes were removed. The treatment was carried out twice a day for three days in addition to the normal analgesic and antibiotics drugs taken by the patient. After the last treatment session, VAS and Oxford hip score was re-administered to ascertain their pain intensity and hip disability level.

For the group with no intervention The VAS and Oxford hip score was administered on the first day of contact to ascertain pain intensity and hip disability level . The subject continued on the normal analgesics only till the third day and VAS and Oxford hip score was re-administered to ascertain their pain intensity and hip disability level.

ELIGIBILITY:
Inclusion Criteria:

Patients who recently had hip arthroplasty were recruited for this study

Exclusion Criteria:

* Subjects who had surgery but have infected wounds.
* Patients who had deep vein thrombosis post-surgery.
* Patients who had thrombophlebitis post-surgery.

Ages: 40 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2017-12-16 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
VAS. Visual Analogue Scale | 5 days
  a horizontal 100mm scale made of plastic calibrated from left (no pain) to the right (severe pain). Ratings greater 70mm indicates severe pain, 45 -74 indicates moderate pain, 5-54 indicates mild pain and 0 -5 indicates no pain

SECONDARY OUTCOMES:
Oxford hip score | 5 days
  it is a 12-item patient-reported outcome measure designed to assess disability after surgery to the hip. Each item was scored between 0 and 4, with 4 been the best outcome per question producing overall scores running from 0 to 48(48 being the best outcome); > 41 is excellent, 34 - 41 is good,27 -33 as fair, and <27 is poor.

CONTACTS AND LOCATIONS:
Overall Officials: Adesola O Ojoawo, PhD, Principal Investigator — Obafemi Awolowo University, Ile Ife
Locations (1):
- Obafemi Awolowo University, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared with other researchers outside the study because data of patients should be kept confidential for ethical reaseons

REFERENCES:
- [Background] Abu-Amer Y, Darwech I, Clohisy JC. Aseptic loosening of total joint replacements: mechanisms underlying osteolysis and potential therapies. Arthritis Res Ther. 2007;9 Suppl 1(Suppl 1):S6. doi: 10.1186/ar2170. PMID 17634145
- [Background] Ali J, Yaffe CS, Serrette C. The effect of transcutaneous electric nerve stimulation on postoperative pain and pulmonary function. Surgery. 1981 Apr;89(4):507-12. PMID 6970995
- [Background] Almeida TF, Roizenblatt S, Tufik S. Afferent pain pathways: a neuroanatomical review. Brain Res. 2004 Mar 12;1000(1-2):40-56. doi: 10.1016/j.brainres.2003.10.073. PMID 15053950